CLINICAL TRIAL: NCT07163663
Title: Effectiveness of a HIFT Training Program on Cognitive and Functional Performance in People With Parkinson's Disease
Brief Title: HIFT Training in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Aguilar, Assistant Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 301294
Record Dates: First submitted 2025-08-21; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Neuro-Degenerative Disease

STUDY DESIGN:
Intervention Model Description: The people who will participate in the study will be randomly divided into two groups: experimental group (EG) and control group (CG). The experimental group will carry out a HIFT training program and the control group will follow their physical and cognitive exercise routine, which will be recorded for their control.
Who Masked: Outcomes Assessor
Masking Description: Randomization will be performed using an Excel spreadsheet, following random number filters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group followed their routine of both physical and cognitive exercises that were recorded for their control. Balance exercises, strength and aerobic exercise. They were assessed at the beginning and at the end of the 10 weeks.
  Interventions: Other: Hight intensity functional trainning
- HIFT group (Experimental): High-intensity functional training was carried out for 10 weeks. The rehabilitation pillar was based on high-intensity functional training. 45-minute sessions divided into 5 minutes of warm-up, 35 minutes of functional exercises, and 5 minutes of going back to bed and cooling down. The 35 minutes of exercises were divided into 3 categories: lower extremity exercises, upper extremity exercises, and static and dynamic balance and coordination exercises. Each category consists of 3 exercises per session, performing 2 sets with a maximum of 10-RM repetitions. Load progression was progressively increased at weeks 3, 5, and 8 between 40-60% of the 1-RM.
  Interventions: Other: Hight intensity functional trainning

INTERVENTIONS:
Other: Hight intensity functional trainning — Warm-up phase: Low-intensity walking 30-50% MHR combined with dynamic mobility exercises
  High Intensity Functional Training (HIFT)
  The raised HIFT intervention proposal is divided into three exercises:
  1. Strength exercise of the lower limbs such as Sit to Stand / Stand to sit and elevation of the upper limbs up in a standing position or lateral gait with knee flexion of one limb among many others.
  2. Upper limb strength exercises: In a standing position with a medicine ball and in front of the wall, throw the ball against it and catch it o Walk while taking the medicine ball from right to left with smooth rotation of the trunk among many others.
  3. Coordination and balance exercises: Go up and down stairs or steps in four steps with arms stretched out in front of you and exercises such as standing, knee flexion and raising the contralateral hand with weights.
  Cooling phase: Stretching of upper and lower limb muscle groups and head and neck muscles.

SUMMARY:
Parkinson's disease (PD) is a progressive and chronic neurodegenerative disease, which presents signs and symptoms both motor (impaired gait, posture, balance, etc.) and cognitive (memory loss, dementia, etc.), all of which cause disability and assuming a high economic cost. Currently, there are already certain authors who have shown how a high-intensity interval training (HIIT) protocol produces improvements in cognitive and physical performance in healthy adults and in people with multiple sclerosis. However, another modality has been created, such as high-intensity functional training (HIFT), which can benefit different populations, both healthy and pathological, due to the multimodal nature of the exercises. These are prescribed knowing the target group and involve the whole body using universal motor recruitment patterns in multiple planes of movement such as squats. The main hypothesis of the study is that high-intensity functional training (HIFT), at a motor and cognitive level, provides a greater benefit than conventional programs of strength, balance and cognition, on the functionality and cognitive capacity of people with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive and chronic neurodegenerative disease, which presents signs and symptoms both motor (impaired gait, posture, balance, etc.) and cognitive (memory loss, dementia, etc.), all of which are causing disability and assuming a high economic cost.

This pathology is characterized by the destruction, due to still unknown causes, of the dopaminergic neurons, which are found in a region of the brain called the basal ganglia, specifically in a part of the brainstem called the substantia nigra. These neurons act in the central nervous system and use dopamine as their primary neurotransmitter, responsible for transmitting the necessary information for the correct control of movements. For this reason, the result of its destruction involves slowing of movements along with lack of coordination.

These processes cause multiple deficits in higher cortical functions, affecting the motor and cognitive capacity of the individual and, therefore, negatively affecting the execution of both basic and instrumental daily activities.

PD is the second most common neurodegenerative disease after Alzheimer's and it presents in both sexes in a similar way, with a slight predominance in men. The World Health Organization already estimated in 2005 a global incidence of 4.5-19 new cases per year per 100,000 inhabitants and a global prevalence of 100-200 cases per 100,000 inhabitants, while a more recent report published by the European Parkinson's Disease Association estimates a worldwide prevalence for the year 2030 of between 8.7 and 9.3 million people. 70% of patients are people over 65 years of age, and 15% of all those affected are adults under 45 years of age. As a general rule, PD affects 1% of the population over 60 years of age, 2% of those over 70 years of age, and 3% of those over 803.

Due to all the physical and psychological consequences that can occur, the economic impact of this type of neurodegenerative pathology in the family nucleus is really great. The average annual expenditure per family unit for the different neurological pathologies is 13,063 euros. If the investigators focus on the EP, the amount is established up to the figure of 9,219 euros per year. This expense is usually progressive according to the degree of advancement of the disease, averaging an expense of 7,146 euros in the incipient phase of the disease, going through 8,491 euros in the intermediate phase and reaching 14,443 euros in the advanced phase. From all this it can be deduced that families are currently the main providers of support services for this type of patient, causing a very high cost for them. In this sense, it is important to highlight that a large percentage of patients have had to change their address or have had to carry out reforms to adapt the home to their situation (bathroom, adjustable bed, crane, restraints or barriers for the bed, among others).

Currently, there are already certain authors who have shown how a high-intensity interval training (HIIT) protocol produces improvements in cognitive and physical performance in healthy adults6 and in people with multiple sclerosis 7,8. These training programs are of a unimodal nature, that is, specific exercises for a specific joint and muscle group such as jumping, rowing, running or lifting weights, among others. However, another modality has been created, such as high-intensity functional training (HIFT), which can benefit different populations, both healthy and pathological, due to the multimodal nature of the exercises. These are prescribed knowing the target group and involve the whole body using universal motor recruitment patterns in multiple planes of movement such as squats. Thanks to multimodality, more aspects such as agility, coordination and precision of movements are worked on compared to unimodal HIIT programs that make this relevant work difficult in a person's daily life. However, the functionality of the exercises provides added value, since it improves the motivational factor, which in turn increases adherence to the program9 and the obtaining of health benefits.

The current study aims to demonstrate the effectiveness of a HIFT training protocol in a specific population, such as people with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease.
2. Phase I or II (Hoehn - Yahr Scale).
3. Independent ambulation for 10 consecutive minutes.
4. Perform physical exercise on a regular basis.

Exclusion Criteria:

1. Medical contraindication for physical activity, deafness or limited hearing and very low vision or blind.
2. Vestibular disorders that compromise balance.
3. Serious psychotic or cognitive disorder.
4. Decompensation or changes in medication.
5. Surgical intervention in the last 6 months.
6. Sedentary people

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Sociodemographic and neurological data registration form | At week 0
  Form for registering clinical history, sociodemographic data and neurological history of each participant, as well as personal and contact information.
Short Form 12-item Questionnaire | At week 0 and 11
  Short Form 12-item Questionnaire is a generic health-related quality of life measurement instrument. It was born as an abbreviated version of the Short Form 36-item Questionnaire, since it consists of 12 items compared to the 36 items of the original and its administration time is approximately 2 minutes. The measurement is based on a Likert-type dichotomous scale, with a different number of response categories, between three and six. The scores of the twelve items were standardized to later place them in a range between 0 and 100. The objective is to evaluate the degree of well-being and functional capacity of people over 14 years of age. This test includes 2 dimensions that represent 8 health concepts most frequently used when measuring quality of life, as well as aspects related to illness. The higher the score, the healthier the person is.
Barthel index | At week 0 and 11
  It was first described by Mahoney and Barthel in 1965 and is widely used by clinicians and researchers. The BI is defined as a generic measure that assesses the patient's level of independence with respect to performing some activities of daily living (ADL), through which different scores and weights are assigned according to the ability of the examined subject to carry out carry out these activities. The values assigned to each activity are based on the time and amount of physical assistance required if the patient is unable to perform that activity. It is made up of ten basic activities that include feeding, dressing and undressing, washing, using the toilet, urination control, stool control, transfers, use of personal hygiene, going up and down stairs and walking. The scores range from 0 to 10 points, passing through 5. 0 is totally dependent on the third person, 5 means that he needs some help and 10 is totally independent.
Short physical performance battery (SSPB) | At week 0 and 11
  The test includes 3 spheres as described below:
  1. Balance test A. Stand with feet together side by side B. Semi-tandem C. Full tandem
  2. Walking speed test: Walk 4 meters and record the time.
  3. Chair rise test: Sit down and get up from the chair 5 times and record the time spent.
  Each test is scored from 0 to 4. The total score ranges from 0 to 12 points.
Fall Risk Assessment Score Scale | At week 0 and 11
  The Fall Risk Assessment Score Scale is a tool that was developed to predict the risk of falls in older people. It is based on five questions about the last year: history of falls in the last 12 months (2 points); decreased gait or noticeable changes in it (1.5 points); loss of balance in the last 12 months (1 point); visual deficit (1 point); decreased grip strength in the hands (1 point). Each variable is associated with a different score, indicated in parentheses at the end of each item. The final score of the scale varies between 0 and 6.5, in such a way that the higher the score, the greater the probability of suffering a fall. Thus, the cut-off value for this scale is 3.5 points, by which scores higher than this are considered to imply risk of falls.
2 minute walk test (2-MWT) | At week 0 and 11
  The 2-MWT15 is a simple, inexpensive, and easy-to-administer test that consists of measuring the maximum distance that the patient is able to walk in 2 minutes, in a short walk in a corridor, simultaneously evaluating the heart rate, the saturation of oxygen and the degree of dyspnea using the Borg scale. Its physiological basis is that the distance achieved on a flat course during the defined time (2 minutes) is an expression of the individual's capacity for submaximal exercise, which allows an evaluation of this capacity in different respiratory pathologies. The 2-MWT influences, in addition to an underlying cardio-respiratory pathology, motivational and musculoskeletal factors that provide a global assessment of exercise capacity and can reflect the daily activity of patients better than other laboratory tests.
Mini Mental State Examination | At week 0 and 11
  It is a brief test that assesses cognitive function. The questions included in the test attempt to examine various areas of cognitive function: orientation, registration, concentration, memory, language, and copying a figure. The Mini Mental State Examination total score is widely accepted as an indicator of the severity of cognitive impairment. Sensitivity is 87% and specificity is 82% in detecting dementia. Likewise, the values obtained in test-retest, 0.89, and from the inter-rater, 0.82, have also shown that Mini Mental State Examination is an effective instrument in the English language. Concurrent validity has been tested with extensive neuropsychological tests and also in longitudinal studies.
  The test has been widely used in clinical practice and in research.
Trail Making Test A y B | At week 0 and 11.
  The test with part A and B measures visual search, scanning, processing speed, mental flexibility and executive functions. In Part A, the subject uses a pencil to connect a series of 25 circled numbers in numerical order on a sheet of paper with the prompt to do so in the shortest time possible. This makes it possible to accurately measure search tools and visual attention and psychomotor speed. In part B, a similar execution is required, with the exception that the person must alternate the sequence of numbers from 1 to 13 with letters from "A" to "L". In this way, we can obtain data on executive control, cognitive flexibility and alternation. The evaluated person is timed, obtaining the resulting time. If the examiner notices an error in the order of the lines drawn, she must interrupt the subject and correct the error without stopping the stopwatch during the correction.
Borg scale | For 10 weeks
  It is a standardized and validated visual analog scale in Spanish, quick and easy to apply, which allows graphically evaluating the subjective perception of respiratory distress or physical effort exerted. The Borg scale has been used since the 1970s and the modified one since the 1980s, which has a range from 0 to 10. The scale determines the intensity of dyspnea and has a written expression added to the number, which helps to categorize the sensation of dyspnea of the subject to whom the test is performed. The result is recorded and coded. The interval between the ranges of the scale increases progressively, number 10 shows the greatest perception of dyspnea (of effort). The modified Borg scale is easy to use if the patient is properly instructed.

CONTACTS AND LOCATIONS:
Overall Officials: MARTA AGUILAR, Study Director — PROFESSOR DOCTOR
Locations (2):
- Spain (2):
  - Ismael Vargas Villanueva, Ibiza Town, Balearic Islands
  - Ismael Vargas Villanueva, Elche, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan WLS, Pin TW. Reliability, validity and minimal detectable change of 2-minute walk test, 6-minute walk test and 10-meter walk test in frail older adults with dementia. Exp Gerontol. 2019 Jan;115:9-18. doi: 10.1016/j.exger.2018.11.001. Epub 2018 Nov 10. PMID 30423359
- [Background] Campbell E, Coulter EH, Paul L. High intensity interval training for people with multiple sclerosis: A systematic review. Mult Scler Relat Disord. 2018 Aug;24:55-63. doi: 10.1016/j.msard.2018.06.005. Epub 2018 Jun 13. PMID 29936326
- [Background] de Lau LM, Breteler MM. Epidemiology of Parkinson's disease. Lancet Neurol. 2006 Jun;5(6):525-35. doi: 10.1016/S1474-4422(06)70471-9. PMID 16713924
- [Background] Wens I, Dalgas U, Vandenabeele F, Grevendonk L, Verboven K, Hansen D, Eijnde BO. High Intensity Exercise in Multiple Sclerosis: Effects on Muscle Contractile Characteristics and Exercise Capacity, a Randomised Controlled Trial. PLoS One. 2015 Sep 29;10(9):e0133697. doi: 10.1371/journal.pone.0133697. eCollection 2015. PMID 26418222
- [Background] Coetsee C, Terblanche E. The effect of three different exercise training modalities on cognitive and physical function in a healthy older population. Eur Rev Aging Phys Act. 2017 Aug 10;14:13. doi: 10.1186/s11556-017-0183-5. eCollection 2017. PMID 28811842
- [Background] Weintraub D, Moberg PJ, Duda JE, Katz IR, Stern MB. Effect of psychiatric and other nonmotor symptoms on disability in Parkinson's disease. J Am Geriatr Soc. 2004 May;52(5):784-8. doi: 10.1111/j.1532-5415.2004.52219.x. PMID 15086662
- See also: Reference values of the Short Physical Performance Battery for patients aged 70 and over in primary health care — http://www.clinicalkey.es